CLINICAL TRIAL: NCT01834443
Title: Therapeutic Effects of Galvanic Vestibular Stimulation (GVS) on Spatial Neglect
Acronym: GVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Schoen Clinic Bad Aibling (Other)
Collaborators: German Center for Vertigo and Balance Disorders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GVS-Therapy
Record Dates: First submitted 2013-04-03; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Spatial Neglect After Right Brain-damage
Keywords: spatial neglect; galvanic vestibular stimulation as therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GVS CL (Experimental): Transmastoid galvanic vestibular stimulation is applied, with the cathode placed on the left mastoid
  Interventions: Device: Direct current galvanic vestibular stimulation
- GVS CR (Experimental): Transmastoid galvanic vestibular stimulation is applied, with the cathode placed on the right mastoid
  Interventions: Device: Direct current galvanic vestibular stimulation
- GVS Sham (Sham Comparator): Transmastoid galvanic stimulation set-up is applied, with only 30s of stimulation
  Interventions: Device: Direct current galvanic vestibular stimulation

INTERVENTIONS:
Device: Direct current galvanic vestibular stimulation
  Other Names: Eldith DC-stimulator manufactured by neuroconn; Model-no 0008; Serial-no 0028

SUMMARY:
The purpose of this study is to determine whether galvanic vestibular stimulation is effective in the treatment of spatial neglect after right brain-damage.

ELIGIBILITY:
Inclusion Criteria:

* spatial neglect after unilateral ischemic infarction or unilateral haemorrhage

Exclusion Criteria:

* Chronic epilepsy
* Metallic implants (including pacemakers)
* Brain tumors
* Scalp inflammation
* Degenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Change in Neglect Test (NET)due to intervention, the German version of the Behavioral Inattention Test (BIT) | Baseline, Post (day after last intervention session), Follow-up 1 (2 weeks after post testing), Follow-up 2 (4 after post testing)

SECONDARY OUTCOMES:
Change in visual-tactile search task due to intervention | Baseline, Post (day after last intervention session), Follow-up 1 (2 weeks after post testing), Follow-up 2 (4 after post testing)
  Subjects searches objects glued to a board, the time needed to do so is measured
Change in subjective haptic vertical due to intervention | Baseline, Post (day after last intervention session), Follow-up 1 (2 weeks after post testing), Follow-up 2 (4 after post testing)
  The haptic vertical is assessed with a wooden device, where subjects are asked to adjust a rod into a vertical position. Deviations (in degrees) are measured.

OTHER OUTCOMES:
Change in subjective visual vertical due to intervention | Baseline, Post (day after last intervention session), Follow-up 1 (2 weeks after post testing), Follow-up 2 (4 after post testing)
  The visual vertical is assessed with the bucket test, in which subjects are asked to indicate when a visual line is vertical for them. Deviations (in degrees) are measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Schoen Clinic Bad Aibling, Bad Aibling, Bavaria, Germany